CLINICAL TRIAL: NCT01246362
Title: A Randomized Controlled Trial to Study the Efficacy of Pre-emptive Etoricoxib in Reducing Postoperative Pain and Improving Functional Outcome in Total Knee Arthroplasty
Brief Title: Efficacy Study of Pre-emptive Etoricoxib for Postoperative Pain and Functional Outcome in Total Knee Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACL-3
Record Dates: First submitted 2010-11-21; First posted 2010-11-23 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Given placebo tablets preoperatively
  Interventions: Drug: Control
- Etoricoxib (Active Comparator): Given etoricoxib preoperatively
  Interventions: Drug: Etoricoxib

INTERVENTIONS:
Drug: Control — Given placebo
  Arms: Control
Drug: Etoricoxib — Given etoricoxib 120mg 24 hours preoperatively and 120mg 2 hours preoperatively
  Arms: Etoricoxib

SUMMARY:
The purpose of this study is to study the efficacy of pre-emptive etoricoxib in reducing post-operative pain and improving function outcome after a total knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most commonly performed orthopaedic surgeries worldwide and has proven to be a success in the treatment of end-stage osteoarthritic knees. TKA is associated with significant postoperative pain which may delay the patient's functional recovery and necessitate an increased use of opioid analgesias, which are themselves associated with significant adverse effects such as nausea and vomiting. The selective cycloxygenase (COX)-2 inhibitor rofecoxib was previously shown in a clinical trial in a paper by Buvanendran et al to reduce postoperative opioid requirement and improve clinical outcomes. Feng et al studied the use of a single dose of rofecoxib pre-operatively and its effect on inflammatory markers and postoperative pain. Rofecoxib has, however, been withdrawn from the market due to its association with cardiovascular side effects. Our current clinical practice in post-operative pain management constitutes post-operative etoricoxib but we hypothesize that pre-emptively administering etoricoxib pre-operatively would give an even greater benefit in terms of post-operative opioid usage, pain scores, and functional recovery in the first 2-3 days. To date, there has been no study investigating etoricoxib as a pre-emptive medication in patients undergoing total knee arthroplasty. We aim to conduct a study to test the efficacy of pre-emptive etoricoxib in reducing postoperative pain, opioid requirement and improving the rate of functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 50 and 80 who are listed for single-knee TKA at Singapore General Hospital by one of 4 adult reconstructive surgeons for the treatment of osteoarthritis will be recruited upon the patient giving written informed consent.

Exclusion Criteria:

* - Younger than 50, older than 80
* Known allergy to etoricoxib or other cycloxygenase-2 inhibitors, aspirin or any Non-steroidal Anti-inflammatory Drugs (NSAIDs)
* American Society of Anaesthesiologists (ASA) grade IV
* Renal insufficiency (Creatinine > 110)
* Known coagulation or hepatic disorder
* Inflammatory arthritis
* Inflammatory bowel disease
* Concurrent conditions which would affect interpretation of pain eg spinal stenosis, lumbar nerve root impingement
* Depression or usage of opioids, sedatives or hypnotics preoperatively
* Special classes of subjects including those pregnant, cognitively impaired, prisoners or institutionalized patients
* Patients with clinically significant abnormalities of laboratory safety tests at baseline, or a history of significant clinical or laboratory abnormality that in the opinion of the investigator would contraindicate the use of etoricoxib
* Patients with unstable hypertension, uncontrolled diabetes mellitus, New York Heart Association (NYHA) class II-IV congestive heart failure, ischaemic heart disease, cerebrovascular disease or peripheral vascular disease (including patients who have recently undergone coronary artery bypass graft of angioplasty)
* Patients with active gastric ulceration or gastrointestinal bleeding
* Patients with a history of any illness that in the opinion of the investigator may confound the results of the study or pose additional risks to the patient
* Occurrence of any surgical complication would exclude the patient from analysis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-07; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Within first 5 days after operation
Functional recovery postoperatively | Within first 5 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Shi-lu Chia, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore